CLINICAL TRIAL: NCT04504344
Title: Non-invasive Brain Stimulation to Improve Quadriceps Muscle Function After Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcadia University (Other)
Responsible Party: Principal Investigator, Ryan Zarzycki, Assistant Professor Department of Physical Therapy, Arcadia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NC NM4R Pilot Project Program
Record Dates: First submitted 2020-07-20; First posted 2020-08-07 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Quadriceps Muscle Weakness; Transcranial Direct Current Stimulation
Keywords: corticospinal excitability
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Active tDCS
  Interventions: Device: Anodal transcranial direct current stimulation (tDCS) - Soterix Medical Inc, 1x1 tDCS (conventional)
- Sham tDCS (Sham Comparator): Sham tDCS
  Interventions: Device: Anodal transcranial direct current stimulation (tDCS) - Soterix Medical Inc, 1x1 tDCS (conventional)

INTERVENTIONS:
Device: Anodal transcranial direct current stimulation (tDCS) - Soterix Medical Inc, 1x1 tDCS (conventional) — We will compare the effects of active versus sham tDCS on quadriceps strength and corticospinal excitability in patients recovering from ACLR.

SUMMARY:
Quadriceps muscle dysfunction persists for years after anterior cruciate ligament reconstruction (ACLR) and is related to poor self-reported outcomes, altered movement patterns and joint loading associated with post-traumatic knee osteoarthritis (OA), and higher risk of reinjury. Emerging evidence indicates that central drive (pathway from the brain to the muscle of interest, i.e corticospinal excitability) to the quadriceps muscle is reduced as early as 2 weeks after surgery and can persist for years after ACLR, meaning that current rehabilitation strategies may not be addressing potential maladaptive changes in central drive. Anodal tDCS is a neurostimulation technology that increases brain excitability (i.e. central drive) and has the potential to address alterations in central drive and quadriceps muscle performance. The purpose of this study is twofold: 1) to determine the effects of anodal tDCS on central drive and quadriceps muscle performance in patients after ACLR, and 2) determine the relationship between central drive and quadriceps muscle performance in patients after ACLR. Central drive will be defined by two measures: 1) active motor thresholds, and 2) slope of a stimulus response curve. Quadriceps muscle performance will be defined by two measures: 1) isometric quadriceps strength, and 2) rate of torque development (RTD). For purpose 1 the investigators hypothesize that measures of central drive and quadriceps muscle performance will increase with administration of active anodal tDCS compared to no change with sham tDCS. For purpose 2 the investigators hypothesize that both measures of central drive will be associated with both measures of quadriceps performance, with a stronger association between central drive and RTD. Following a cross-over design patients 3-6 months from ACLR will receive active and sham anodal tDCS at different sessions separated by 7-10 days while they ride a stationary bike for 20 minutes. Bike position and intensity will be standardized for all patients to maximize quadriceps activity. Findings from this study will expand our basic science knowledge on how tDCS effects different aspects of corticospinal excitability and quadriceps strength, and lead to subsequent studies to determine the effects of multiple sessions of tDCS on corticospinal excitability and quadriceps muscle performance in patients recovering from ACLR.

ELIGIBILITY:
Inclusion Criteria:

-Underwent primary ACL reconstruction within 3-6 months

Exclusion Criteria include:

* multiple ligament reconstruction
* osteo-chondral procedures
* any previous lower extremity surgery
* previous ACL injury
* Metal or implants in the head or neck
* history of neurological disease, seizures, severe migraines, and concussion within the last 6 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
isometric quadriceps torque | 3-6 months after ACL Reconstruction
  Nm
quadriceps rate of torque development | 3-6 months after ACL Reconstruction
  Nm/s
Corticospinal excitability - active motor threshold | 3-6 months after ACL Reconstruction
  percent maximal stimulator output
Corticospinal excitability - slope of the stimulus response curve | 3-6 months after ACL Reconstruction
  motor evoked potential/percent active motor threshold

CONTACTS AND LOCATIONS:
Locations (1):
- Ryan Zarzycki, Glenside, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zarzycki R, Leung A, Abraham R, Hammoud S, Perrone M, Kantak S. Determining the safety, feasibility, and effects of anodal transcranial direct current stimulation on corticospinal excitability and quadriceps performance after anterior cruciate ligament reconstruction: a randomized crossover design. Ann Jt. 2025 Jan 21;10:3. doi: 10.21037/aoj-24-15. eCollection 2025. PMID 39981427
- [Derived] Leung A, Kantak S, Hammoud S, Abraham R, Zarzycki R. Sex differences in corticospinal excitability and quadriceps performance after anterior cruciate ligament reconstruction. J Orthop Res. 2024 Apr;42(4):769-776. doi: 10.1002/jor.25725. Epub 2023 Nov 27. PMID 37938095

DOCUMENTS (2):
  • Study Protocol (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT04504344/Prot_001.pdf
  • Informed Consent Form (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT04504344/ICF_000.pdf